CLINICAL TRIAL: NCT02732665
Title: Sensitivity and Specificity of Glycosaminoglycan Scores in the Diagnosis of Early Progression in Advanced Renal Cell Carcinoma
Brief Title: Glycosaminoglycan Scores as Monitoring Biomarkers in Advanced Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Jens Nielsen (Other)
Collaborators: Sahlgrenska University Hospital (Other); University of Modena and Reggio Emilia (Other)
Responsible Party: Sponsor-Investigator, Jens Nielsen, Professor, Chalmers University of Technology
Organization: Chalmers University of Technology (Other)
Other Study IDs: GAG-RCC-02
Record Dates: First submitted 2016-03-16; First posted 2016-04-11 (Estimated); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ethylenediaminetetraacetic acid (EDTA)-plasma from blood obtained through venipuncture; and any-void urine.
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, glycosaminoglycan (GAG) profiling in subjects diagnosed with metastatic renal cell carcinoma (mRCC) is hypothesized to be useful in monitoring drug response and predict radiological response. To this end, glycosaminoglycan scores based on longitudinal samples of plasma and urine in prospectively enrolled patients will be correlated to radiological response to first-line therapy based on current standard-of-care. A positive correlation indicates that glycosaminoglycan scores can successfully detect patients that are not responding to treatment before the scheduled follow-up in which radiological imaging is performed. Data on the extent of metastasis (number of metastatic sites) will be collected to assess whether glycosaminoglycans correlate accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Diagnosis of renal cell carcinoma
* Metastatic disease
* Predicted life expectancy over 2 months
* Patient referred for first line drug therapy
* Standard imaging evaluation 12 weeks prior to inclusion
* Planned for standard imaging within 16 weeks after start of therapy
* Informed consent

Exclusion Criteria:

* Lack of proper compliance to accept continuous samplings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Untreated patients with diagnosis of metastatic renal cell carcinoma referred for first line treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic (ROC) curve (AUC) for the sensitivity/specificity of plasma/urine glycosaminoglycan scores to progressive disease at response evaluation | 6 weeks and every 3 months after treatment start up to 12 months
  ROC curves are generated to determine the specificity and sensitivity of the glycosaminoglycan scores sampled at 6 weeks and every 3 months to progressive disease as assessed by radiological imaging during the scheduled response evaluation according to RECIST 1.1. criteria. The area under each ROC curve (AUC) is then calculated as primary outcome measure.

SECONDARY OUTCOMES:
Area under the receiver operating characteristic (ROC) curve (AUC) for the sensitivity/specificity of plasma/urine glycosaminoglycan scores in early prediction of objective response at first response evaluation | Baseline; 6 weeks after treatment start
  ROC curves are generated to determine the specificity and sensitivity of the glycosaminoglycan scores sampled at 6 weeks to complete response or partial response as assessed by radiological imaging during the first scheduled response evaluation according to RECIST 1.1. criteria. The area under each ROC curve (AUC) is then calculated as primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Nielsen, PhD, Principal Investigator — Chalmers University of Technology; Ulrika Stierner, M.D. PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data will be accessible upon study publication

REFERENCES:
- [Result] Gatto F, Bratulic S, Jonasch E, Limeta A, Maccari F, Galeotti F, Volpi N, Lundstam S, Nielsen J, Stierner U. Plasma and Urine Free Glycosaminoglycans as Monitoring and Predictive Biomarkers in Metastatic Renal Cell Carcinoma: A Prospective Cohort Study. JCO Precis Oncol. 2023 Feb;7:e2200361. doi: 10.1200/PO.22.00361. PMID 36848607